CLINICAL TRIAL: NCT04649567
Title: COLONIC RESECTION FOR CANCER AS DIABETOGENIC RISK FACTOR - A Study of the Pathophysiological Effects of Colon Resection on Glucose Homeostasis
Brief Title: COLONIC RESECTION FOR CANCER AS DIABETOGENIC RISK FACTOR
Acronym: COLECDIAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Herlev Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Maria Saur Svane, Investigator, Hvidovre University Hospital
Other Study IDs: H-20015184
Record Dates: First submitted 2020-09-02; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Glucose Metabolism Disorders; Colon Cancer; Surgery; Chemotherapy Effect
MeSH Terms: conditions — Glucose Metabolism Disorders; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colon cancer (CC) survivors have an increased risk of developing T2D. A recent study revealed that the surgical procedures per se may be causally involved. Hence, left-sided colon resections increased the risk of developing T2D. In addition, treatment with chemotherapy may play a role in the pathogenesis. Given the steadily improving survival rate after a CC diagnosis, prevention of secondary diseases such as T2D is important to improve quality of life in these patients and to reduce socioeconomic expenses. This study aims to elucidate the effect of resection of tumors located in the left part of the colon on pathophysiological intermediates, which may lead to T2D 12 months post-surgery or later. The physiological mechanism might be a changed postprandial secretion of gut hormones including glucagon-like peptide-1 (GLP-1) secreted from L-cells in the left part of the colon. The investigators will evaluate changes in primarily glucose homeostasis as well as in gastrointestinal hormones, microbiota, visceral fat accumulation and markers of low-grade inflammation etc. in CC survivors who underwent a left hemicolectomy or sigmoidectomy.

Material and Methods: 60 patients will be included in this explorative clinical study. Patients will be divided into 4 groups depending on surgical procedure and treatment with chemotherapy. In the group of patients undergoing left hemicolectomy or sigmoidectomy ± treatment with chemotherapy 2 x 15 patients will be included, and in the group of patients scheduled to undergo right hemicolectomy ± treatment with chemotherapy another 2 x 15 patients will be included. During the 3 study visits (before surgery, 3-4 weeks post-surgery and 12 months post-surgery) the following tests will be performed: An oral glucose tolerance test, blood and fecal sampling, a DXA scan and an ad libitum meal test.

Implications: With this study the investigators expect to obtain an insight in the pathogenesis behind the possible development of T2D in CC survivors who underwent a resection of the left part of the colon ± treatment with chemotherapy. This insight may also help scientists develop new ways of treating or preventing T2D in general.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

* Adult (> 18 yrs.)
* ASA score 1-3
* Signed written informed consent
* Hba1c <48 mmol/mol
* Hemoglobin ≥ 6,5 mmol/L

Exclusion Criteria:

* • Pregnancy

  * Known type 1 or 2 diabetes
  * Inflammatory bowel disease (Ulcerous colitis and Crohns' disease).
  * Prior major abdominal surgery including bariatric surgery or colorectal resections
  * Treatment with agents that may interfere with glucose homeostasis and or appetite or reduce the chance of successful follow-up examination
  * Planned stoma

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 60 patients diagnosed with colon cancer will be investigated. They have to be planned for surgical resection of a segment of colon (left hemicolectomy, sigmoidectomy or right hemicolectomy) for cancer without signs of metastases (cT1-4N0-2M0), with and without planned treatment with adjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in 2-hour blood glucose (OGTT) 12 months after hemicolectomy ± chemotherapy | 3-4 weeks and 1 year after anticancer treatment

SECONDARY OUTCOMES:
Changes in blood glucose (iAUC) and (tAUC) in response to a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in hemoglobin a1c (HbA1c) | 3-4 weeks and 1 year after anticancer treatment
Changes in fasting blood glucose levels (mmol/L) | 3-4 weeks and 1 year after anticancer treatment

OTHER OUTCOMES:
changes in GLP-1 (iAUC) to a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
changes in bacterial composition in fecal samples | 3-4 weeks and 1 year after anticancer treatment
changes in appetite during an ad libitum meal test by VAS scale (1-10). 10 represents highest value. | 3-4 weeks and 1 year after anticancer treatment
Changes in body weight | 3-4 weeks and 1 year after anticancer treatment
Changes in body composition (fat, bone and lean tissue) by DXA scan | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of leucocytes | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of neutrophils | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of hs-CRP | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of IL-6 | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of soluble IL-6 receptor | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of IL-1Ra | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of INF-γ | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of TNF-α | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of leptin | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of adiponectin | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of IL-10 | 3-4 weeks and 1 year after anticancer treatment
changes in plasma concentration of IL-8 | 3-4 weeks and 1 year after anticancer treatment
Changes in fasting plasma bile acids concentrations | 3-4 weeks and 1 year after anticancer treatment
Changes in gastric emptying rate by plasma paracetamol concentrations during a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in systemic lipid concentration by fasting plasma triglycerides, HDL and LDL cholesterol | 3-4 weeks and 1 year after anticancer treatment
Changes in unbiased mass-spectrometry (plasma proteomics that captures over 400 circulating proteins in blood including markers of low-grade inflammation and lipid metabolism) | 3-4 weeks and 1 year after anticancer treatment
changes in the metabolome (concentrations of aminoacids) in plasma samples | 3-4 weeks and 1 year after anticancer treatment
changes in the metabolome (concentrations of bile acids) in plasma samples | 3-4 weeks and 1 year after anticancer treatment
changes in the metabolome (concentrations lipids) in plasma samples | 3-4 weeks and 1 year after anticancer treatment
Changes in gene Risk Score for T2D by analysing buffy coat suspension | 3-4 weeks and 1 year after anticancer treatment
Changes in quality of life measured by the questionnaire Functional Assessment of Cancer Therapy (FACT-C) | 3-4 weeks and 1 year after anticancer treatment
Changes in insulin secretion rate (ISR) by an OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in insulinogenic index (IGI) by an OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in β-cell glucose sensitivity (β-GS) by an OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in insulin resistance by HOMA analysis (HOMA-IR) by an OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in disposition index by an OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in insulin clearance by an OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in rates of absorption of the ingested glucose by an OGTT | 3-4 weeks and 1 year after anticancer treatment
Change in physical activity level measured by International Physical Activity Questionnaires (IPAQ) questionnaire | 1 year after anticancer treatment
Changes in PYY (iAUC) response to a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in GLP-2 (iAUC) in responses to a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in GIP (iAUC) in responses to a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
changes in ghrelin (iAUC) in responses to a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in CCK (iAUC) in responses to a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
changes in OXM (iAUC) in responses to a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in neurotensin (iAUC) in responses to a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in glicentin (iAUC) in responses to a 3-hour OGTT | 3-4 weeks and 1 year after anticancer treatment
Changes in gene risk Score for T2D using buffy coat analysis | 3-4 weeks and 1 year after anticancer treatment

CONTACTS AND LOCATIONS:
Overall Officials: Louise L Lehrskov, PhD, MD, Principal Investigator — Rigshopitalet
Locations (2):
- Denmark (2):
  - Rigshopitalet, Copenhagen, Please Select
  - Hvidovre Hospital, Hvidovre